CLINICAL TRIAL: NCT04795908
Title: STOP-TIC Study: Strengthening Tourette Treatment OPtions Using TMS to Improve CBIT
Brief Title: Combined CBIT and rTMS to Improve Tourette's Syndrome
Acronym: STOP-TIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202002701-A; OCR40702 (Other: UF OnCore)
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2023-12

CONDITIONS: Tourette Syndrome
Keywords: TMS; Transcranial magnetic stimulation; CBIT; Comprehensive Behavioral Intervention for Tics; Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Active rTMS Group (Experimental): Patients will be seated in a comfortable reclined chair. The neurostimulation protocol will include 1-Hz rTMS over the bilateral SMA at 110% resting motor threshold (RMT). The SMA will be identified as 4 cm anterior to the vertex (Cz in standard 10-20 EEG setup). Each session will consist of 6 trains lasting 5 minutes each (300 pulses per train) with an intertrain interval of 1 minute for a total duration of 35 minutes (1800 pulses). Patients will receive 4 sessions each day on 4 consecutive days for a total of 16 sessions. Daily duration of this study protocol should last approximately 170 minutes including a 10 minute break in between each session.
  Interventions: Device: Transcranial Magnetic Stimulation; Behavioral: Comprehensive behavioral intervention

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — rTMS will be delivered using a MagStim Super Rapid2 TMS therapy system.
Behavioral: Comprehensive behavioral intervention — Patients will receive CBIT with a therapist trained in CBIT. Each session will last about an hour and will be delivered remotely via telemedicine. Sessions will be tailed to the patient's individual needs.

SUMMARY:
The investigator will apply 16 sessions of repetitive transcranial magnetic stimulation (rTMS) over 4 consecutive days for adult patients suffering from Tourette's Syndrome. Following rTMS, patients will undergo 8 sessions of Comprehensive Behavioral Intervention for Tics (CBIT) over 10 weeks via telemedicine. Clinical improvement in tic severity will be the primary outcome measure. Secondary outcome measures including underlying physiological effects will be measured via functional magnetic resonance imaginge (fMRI), high-density electroencephalograhy (HD-EEG), and TMS.

DETAILED DESCRIPTION:
Patients will be randomly assigned to active or sham stimulation, with 10 in each group, followed by 10 weeks of tele-CBIT. Patients will have primary and secondary outcome measures performed at four time points: Baseline (T0), following rTMS (T1), following CBIT (T2), and 1 month later (T3). The rTMS protocol will consist of 6 trains targeted to the supplementary motor area (SMA) lasting 5 minutes each (300 pulses per train) with an intertrain interval of 1 minute for a total duration of 35 minutes (1800 pulses). Patients will receive 4 sessions each day on 4 consecutive days for a total of 16 sessions. Daily duration of this study protocol should last approximately 170 minutes including a 10 minute break in between each session. The sham protocol will be the same except a sham coil will be used instead of an active coil. Following rTMS, patients will undergo 10 weeks of tele-CBIT.

The following outcome measures will be collected at four timepoints (T0, T1, T2, and T3):

Tics will be examined with the standardized Yale Global Tic Severity Scale (YGTSS) and the modified Rush Videotape Tic Rating Scale (mRVTRS), and co-morbid symptoms with the Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Yale-Brown Obsessive Compulsive Scale (Y-BOCS) and Adult ADHD Self-Reports Scale (ASRS). Quality of life will be assessed with the Gilles de la Tourette Syndrome - Quality of Life scale (GTS-QOL).

TMS measures: A single-pulse of TMS will be targeted over the motor cortex to generate a motor evoked potential (MEP), which can be captured on EMG. The rest of the EMG will be analyzed to assess the time between the TMS pulse and the MEP (also known as the latency) and the amount of time muscle activity remains silent following the MEP (also known as the cortical silent period). In a paired-pulse TMS paradigm, a subthreshold pulse will be provided followed by an interstimulus interval and then subsequent delivery of a suprathreshold pulse. When the interstimulus interval is short (1-4 msec), the ratio of MEP amplitudes produced by these two pulses is known as short interval intracortical inhibition (SICI).

fMRI measure: Functional MRI will be used to record Blood Oxygen Level Dependent (BOLD) activity changes in patients at rest.

HD-EEG measure: A 128-electrode cap will be used to assess electrical activity in patients at rest and actively trying to suppress their tics.

ELIGIBILITY:
Inclusion Criteria:

* Any patient diagnosed with Tourette Syndrome > 18 years of age with moderate tic severity.
* Participants will be allowed to continue oral medications that they are taking for TS concurrently but will not be allowed to change their concurrent medication regimen throughout the duration of the study

Exclusion Criteria:

* Presence of metallic objects or neurostimulators in the brain
* Pregnancy
* History of active seizures or epilepsy
* Contraindications to receiving fMRI, such as claustrophobia
* Inability to participate in CBIT due to other underlying cognitive or medical condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Wagle Shukla, MD, Principal Investigator — University of Florida
Locations (1):
- Fixel Neurologic Institute, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active rTMS Group: Patients will be seated in a comfortable reclined chair. The neurostimulation protocol will include 1-Hz rTMS over the bilateral SMA at 110% resting motor threshold (RMT). The SMA will be identified as 4 cm anterior to the vertex (Cz in standard 10-20 EEG setup). Each session will consist of 6 trains lasting 5 minutes each (300 pulses per train) with an intertrain interval of 1 minute for a total duration of 35 minutes (1800 pulses). Patients will receive 4 sessions each day on 4 consecutive days for a total of 16 sessions. Daily duration of this study protocol should last approximately 170 minutes including a 10 minute break in between each session.
  Transcranial Magnetic Stimulation: rTMS will be delivered using a MagStim Super Rapid2 TMS therapy system.
  Comprehensive behavioral intervention: Patients will receive CBIT with a therapist trained in CBIT. Each session will last about an hour and will be delivered remotely via telemedicine. Sessions will be tailed to the patient's individual needs.
  The 3 patients recruited for this study were assigned to this active rTMS group.
Period: Overall Study
Arm/Group | Active rTMS Group
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active rTMS Group
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 24.67 [18 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Tic Severity
Description: Tic severity will be measured with YGTSS. YGTSS is a clinician-rated scale used to assess tic severity, scored out of 100 where a higher score indicates greater tic frequency and severity. It includes a checklist of motor and vocal tics followed by an assessment of the number, frequency, intensity, complexity, and inference of motor tics and phonic tics - scored separately. Each of these dimensions is scored on a 0 to 5 scale. The YGTSS provides three tic severity scores: Total Motor (0 to 25); Total Phonic (0 to 25) and the combined Total Tic Severity Score (0 to 50), as well as a separate Impairment dimension scored from 0 to 50.
Time Frame: Through study completion, an average of 3 months
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Baseline: Patients will be seated in a comfortable reclined chair. The neurostimulation protocol will include 1-Hz rTMS over the bilateral SMA at 110% resting motor threshold (RMT). The SMA will be identified as 4 cm anterior to the vertex (Cz in standard 10-20 EEG setup). Each session will consist of 6 trains lasting 5 minutes each (300 pulses per train) with an intertrain interval of 1 minute for a total duration of 35 minutes (1800 pulses). Patients will receive 4 sessions each day on 4 consecutive days for a total of 16 sessions. Daily duration of this study protocol should last approximately 170 minutes including a 10 minute break in between each session.
  Transcranial Magnetic Stimulation: rTMS will be delivered using a MagStim Super Rapid2 TMS therapy system.
  Comprehensive behavioral intervention: Patients will receive CBIT with a therapist trained in CBIT. Each session will last about an hour and will be delivered remotely via telemedicine. Sessions will be tailed to the patient's individual needs.
- Post-TMS (Approximately 1 Week): Captured following completion of rTMS, approximately 1 week after baseline.
- Post-CBIT (Approximately 11 Weeks): Captured following tele-CBIT intervention, approximately 11 weeks after baseline.
Arm/Group | Baseline | Post-TMS (Approximately 1 Week) | Post-CBIT (Approximately 11 Weeks)
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | 59.3 [50 to 76] | 43.3 [29 to 49] | 37.67 [26 to 48]
Statistical Analysis 1: Comparison: Baseline vs Post-TMS (Approximately 1 Week) vs Post-CBIT (Approximately 11 Weeks); Test type: Non-Inferiority — looking for statistical significant differences between groups; p = 0.1997, ANOVA

2. Secondary Outcome: Modified Rush Videotape Tic Rating Scale (mRVTRS)
Description: This is a tool used by an objective examiner to quantify the severity of a patient's tics by rating the number of body areas affected, motor tic frequency, phonic tic frequency, motor tic severity, and phonic tic severity, each on a 0 through 4 score by watching a video of the patient. Scored out of 20, where a higher score indicates greater tic severity.
Time Frame: Through study completion, an average of 3 months
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Baseline: Prior to TMS
Arm/Group | Baseline | Post-TMS (Approximately 1 Week) | Post-CBIT (Approximately 11 Weeks)
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | 16.5 [13.5 to 19.5] | 12.33 [11 to 15] | 9.5 [6.5 to 13.5]
Statistical Analysis 1: Comparison: Baseline vs Post-TMS (Approximately 1 Week) vs Post-CBIT (Approximately 11 Weeks); Test type: Non-Inferiority — looking for statistical significant differences between groups; p = 0.076, ANOVA

3. Secondary Outcome: Beck Depression Inventory (BDI)
Description: This is a 21-question survey evaluating depression in patients on a 0 to 3 scale. Scored out of 63 points, where a higher score indicates a higher level of depression.
Time Frame: Through study completion, an average of 3 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Baseline | Post-TMS (Approximately 1 Week) | Post-CBIT (Approximately 11 Weeks)
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | 17 [8 to 26] | 12 [7 to 21] | 11.3 [7 to 17]
Statistical Analysis 1: Comparison: Baseline vs Post-TMS (Approximately 1 Week) vs Post-CBIT (Approximately 11 Weeks); Test type: Non-Inferiority — looking for statistically significant differences between groups; p = 0.6228, ANOVA

4. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: This is a 21-question survey evaluation anxiety in patients on a 0 to 3 scale. Out of 63 points, where a higher score indicates a higher level of anxiety.
Time Frame: Through study completion, an average of 3 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Baseline | Post-TMS (Approximately 1 Week) | Post-CBIT (Approximately 11 Weeks)
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | 21.67 [10 to 39] | 17 [8 to 32] | 18 [11 to 29]
Statistical Analysis 1: Comparison: Baseline vs Post-TMS (Approximately 1 Week) vs Post-CBIT (Approximately 11 Weeks); Test type: Non-Inferiority — looking for statistically significant differences between groups; p = 0.8984, ANOVA

5. Secondary Outcome: Yale-Brown Obsessive Compulsive Scale (Y-BOCS)
Description: This is a 10 question survey which rates components of obsessive thoughts or compulsive behavior and each question is rated on a 0 through 4 scale. Scored out of 40, where a higher score indicates higher levels of obsessive-compulsive tendencies.
Time Frame: Through study completion, an average of 3 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Baseline | Post-TMS (Approximately 1 Week) | Post-CBIT (Approximately 11 Weeks)
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | 17 [13 to 21] | 18.3 [12 to 22] | 20 [14 to 28]
Statistical Analysis 1: Comparison: Baseline vs Post-TMS (Approximately 1 Week) vs Post-CBIT (Approximately 11 Weeks); Test type: Non-Inferiority — looking for statistically significant differences between groups; p = 0.8188, ANOVA

6. Secondary Outcome: Adult ADHD Self-Report Scale (ASRS)
Description: This is an 18-question survey which asks patients to rate levels of attention, concentration, and organization as applied to daily tasks. Each question was assigned to a Likert scale of 1-5, where a higher number indicates a higher severity of that aspect of attention deficit. Individual responses were then summed together to obtain a Total Score ranging from 18-90, where a higher score indicates a higher impact of ADHD symptoms on daily functioning.
Time Frame: Through study completion, an average of 3 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Baseline | Post-TMS (Approximately 1 Week) | Post-CBIT (Approximately 11 Weeks)
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | 70.67 [70 to 72] | 64.33 [60 to 68] | 62 [59 to 65]
Statistical Analysis 1: Comparison: Baseline vs Post-TMS (Approximately 1 Week) vs Post-CBIT (Approximately 11 Weeks); Test type: Non-Inferiority — Looking for statistically significant differences between groups; p = 0.0288, ANOVA

7. Secondary Outcome: Gilles de la Tourette Syndrome - Quality of Life Scale (GTS-QOL)
Description: This is a 27-question survey that asks patients to rate how their tics and abnormal movements affect their quality of life. When answers are converted to a Likert value of 1 through 5, the survey is scored out of 135, with higher scores indicating worse quality of life.
Time Frame: Through study completion, an average of 3 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Baseline | Post-TMS (Approximately 1 Week) | Post-CBIT (Approximately 11 Weeks)
Number analyzed (Participants) | 3 | 3 | 3
score on a scale | 87.33 [80 to 100] | 67.67 [60 to 78] | 64.67 [57 to 74]
Statistical Analysis 1: Comparison: Baseline vs Post-TMS (Approximately 1 Week) vs Post-CBIT (Approximately 11 Weeks); Test type: Non-Inferiority — looking for statistically significant differences between groups; p = 0.0524, ANOVA

8. Secondary Outcome: High-Density EEG
Description: High-Density EEG was measured while patients either allowed tics to come or actively suppressed tics
Time Frame: 12 weeks
Population: Unable to be completed due to technical limitations
Arm/Group | Baseline | Post-TMS (Approximately 1 Week) | Post-CBIT (Approximately 11 Weeks)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 11-12 weeks
Groups:
- Post-TMS: follow rTMS
- Post-CBIT: following tele-CBIT
Arm/Group | Baseline | Post-TMS | Post-CBIT
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 3/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline (N=3) | Post-TMS (N=3) | Post-CBIT (N=3)
Headache (Nervous system disorders) | 0 | 3 (3) | 0 — 2 participants had mild transient headaches and 1 participant with a known migraine disorder had a migraine following stimulation with rTMS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT04795908/Prot_SAP_000.pdf